CLINICAL TRIAL: NCT00461734
Title: PROTECT-PACE STUDY - The Protection of Left Ventricular Function During Right Ventricular Pacing. Does Right Ventricular High-septal Pacing Improve Outcome Compared With Right Ventricular Apical Pacing?
Brief Title: PROTECT-PACE STUDY - The Protection of Left Ventricular Function During Right Ventricular Pacing
Acronym: PROTECT-PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROTECT-PACE Version 4
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Left Ventricular Dysfunction
Keywords: Right Ventricular High Septal Pacing; Right Ventricular Apical Pacing; Left Ventricular Dysfunction; Heart Block; Pacemaker; Atrial Fibrillation; Ejection Fraction
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Block; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RV Apex (Active Comparator)
  Interventions: Other: RV lead placement site
- RV High Septum (Experimental)
  Interventions: Other: RV lead placement site

INTERVENTIONS:
Other: RV lead placement site — Patients randomised to RV apical or high septal lead placement site

SUMMARY:
This study will be done in patients who require the implantation of a cardiac pacemaker (an electronic device that controls the heartbeat) for complete heart block (a heart rhythm abnormality resulting in a slow heart beat). Pacemakers regulate the heart beat by delivering pulses of electricity through special wires (pacing leads) which are placed inside the heart.

This study will compare two groups of pacemaker patients. Each group will have their pacing leads placed in a particular location in the heart. The purpose of the study is to show whether the position used in one group is better for maintaining effective heart function compared to the position used in the other group.

The leads in one group will be placed in a position called the Right Ventricular Apex. This is the traditional and most frequently used position for pacemaker leads.

The leads in the other group will be placed in a position called the Right Ventricular High Septum. This is a less commonly used position, but may result in health benefits for the patients compared with the Right Ventricular Apex.

DETAILED DESCRIPTION:
There is an increasing amount of evidence to suggest that other positions in the heart may be more effective than the conventional Right Ventricular Apex (RVA) position for restoring good heart function. The best site to place a lead has not yet been proven.

This is a study comparing the long term clinical effects of two different lead positions. The measurements taken to assess the clinical effects include:

* the effectiveness of the heart's pumping action (as measured by ultrasound scans)
* measurements of how far patients can walk in 6 minutes
* analysis of blood samples
* collection of information from the pacemaker about heart rhythm problems

Half of the patients in the study will receive conventional leads placed in the more common RVA position in the heart. The other half will receive a relatively new type of lead placed in what is called the Right Ventricular High Septal (RVHS) position.

In order to fairly compare the outcomes of these two different lead positions this study has been designed as a 'randomized', 'blind' trial. This means that the group which patients will be entered into will be chosen at random and patients will not be told which group they are in.

Patients will each have an equal (50:50) chance of being in either group. By carefully comparing the clinical differences between the two groups of patients, the study aims to prove whether or not there are additional benefits for patients when the RVHS lead position is used.

All leads used in the study have been shown to be safe for patients and are available commercially for implantation. All of the implanting doctors involved in the study are experienced at implanting the pacemakers and leads that will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high grade AV block and sinus rhythm, scheduled to undergo dual chamber pacemaker implantation OR patients with high grade AV block and permanent atrial fibrillation, scheduled to undergo single chamber ventricular pacemaker implantation.
* Patients aged 18 years or older.

Exclusion Criteria:

* Patients indicated for an Implantable Cardioverter Defibrillator or Cardiac Resynchronization Therapy.
* Patients following junctional ablation.
* Patients with a Myocardial Infarction within three months prior to enrollment.
* Patients that received bypass surgery within three months prior to enrollment.
* Patients that had a valve replacement within three months prior to enrollment or patients with a mechanical right heart valve.
* Patients where a right ventricular lead cannot be placed i.e. complex congenital heart disease.
* Patients with hypertrophic obstructive cardiomyopathy.
* Patients with acute coronary syndrome, unstable angina, severe mitral regurgitation and/or hemodynamically significant aortic stenosis.
* Previous implanted pacemaker or cardioverter defibrillator.
* Known paroxysmal atrial fibrillation or a documented episode of atrial fibrillation prior to enrollment.
* Patients on amiodarone therapy within the last six months prior to enrollment.
* Terminal conditions with a life expectancy of less than two years.
* Participation in any other study that would confound the results of this study.
* Psychological or emotional problems that may interfere with the volunteer's ability to provide full consent or fully understand the purposes of the study.
* Pregnant patients or patients who may become pregnant during the time-scale of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2007-08; Primary Completion 2013-10 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gerald Kaye, Study Chair — Princess Alexandra Hospital
Locations (18):
- Australia (6):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane & Womens' Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Brisbane, Queensland
  - Calvary Wakefield Hospital, Adelaide, South Australia
  - Flinders Medical Center, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
- United Kingdom (10):
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospital of Wales, Cardiff
  - Colchester General, Colchester
  - Leeds General Infirmary, Leeds
  - St. Thomas' Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Norfolk and Norwich University Hospital, Norwich
  - Princess Royal Hospital, Orpington, Kent
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saito M, Iannaccone A, Kaye G, Negishi K, Kosmala W, Marwick TH; PROTECT-PACE investigators. Effect of Right Ventricular Pacing on Right Ventricular Mechanics and Tricuspid Regurgitation in Patients With High-Grade Atrioventricular Block and Sinus Rhythm (from the Protection of Left Ventricular Function During Right Ventricular Pacing Study). Am J Cardiol. 2015 Dec 15;116(12):1875-82. doi: 10.1016/j.amjcard.2015.09.041. Epub 2015 Oct 9. PMID 26517949
- [Derived] Kosmala W, Saito M, Kaye G, Negishi K, Linker N, Gammage M, Marwick TH; Protect-Pace Investigators. Incremental value of left atrial structural and functional characteristics for prediction of atrial fibrillation in patients receiving cardiac pacing. Circ Cardiovasc Imaging. 2015 Apr;8(4):e002942. doi: 10.1161/CIRCIMAGING.114.002942. PMID 25862716
- [Derived] Saito M, Kaye G, Negishi K, Linker N, Gammage M, Kosmala W, Marwick TH; Protect-Pace investigators. Dyssynchrony, contraction efficiency and regional function with apical and non-apical RV pacing. Heart. 2015 Apr;101(8):600-8. doi: 10.1136/heartjnl-2014-306990. Epub 2015 Feb 9. PMID 25666325
- [Derived] Kaye GC, Linker NJ, Marwick TH, Pollock L, Graham L, Pouliot E, Poloniecki J, Gammage M; Protect-Pace trial investigators. Effect of right ventricular pacing lead site on left ventricular function in patients with high-grade atrioventricular block: results of the Protect-Pace study. Eur Heart J. 2015 Apr 7;36(14):856-62. doi: 10.1093/eurheartj/ehu304. Epub 2014 Sep 4. PMID 25189602

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Partecipants initially assessed for eligibility were 248 of whom 8 were excluded before the randomization due to the following causes:
  * 4 failed inclusion/exclusion criteria
  * 2 cheanged medical condition resulting no longer eligible
  * 1 had a non-pacemaker procedure
  * 1 the site was aware of his/her randomization code in the envelope
Groups:
- RV Apex: RV lead placement site: Patients randomised to RV apical lead placement site
- RV High Septum: RV lead placement site: Patients randomised to RV high septal lead placement site
Period: Overall Study
Arm/Group | RV Apex | RV High Septum
Started | 120 | 120
Completed | 62 | 60
Not Completed | 58 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RV Apex | RV High Septum | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 19 | 44
  >=65 years | 95 | 101 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (11.1) | 74.7 (10) | 74.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 32 | 79
  Male | 73 | 88 | 161
Region of Enrollment [Number; unit: participants]
  New Zealand | 12 | 14 | 26
  United Kingdom | 44 | 42 | 86
  Australia | 64 | 64 | 128

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Ejection Fraction From Baseline to 2 Years (Intent to Treat Cohort).
Time Frame: At 2-year follow-up
Population: Intent to Treat Cohort with data available
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- RV Apex: RV lead placement site: Patients randomised to RV apical lead placement site (Intent to treat cohort)
- RV High Septum: RV lead placement site: Patients randomised to RV high septal lead placement site (Intent to treat cohort)
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 88 | 88
percentage | -2.29 (10.5) | -3.43 (8.4)
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.4347, two-sided z-test

2. Primary Outcome: Change in Left Ventricular Ejection Fraction From Baseline to 2 Years (Per Protocol Cohort).
Time Frame: At 2-year follow-up
Population: Per Protocol Cohort with data available
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- RV Apex: RV lead placement site: Patients effectively had RV apical lead placement site (Per protocol cohort)
- RV High Septum: RV lead placement site: Patients effectively had RV high septal lead placement site (Per protocol cohort)
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 89 | 59
percentage | -2.04 (10.4) | -3.60 (7.8)
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.338, two-sided z-test

3. Secondary Outcome: Incidence of Atrial Tachyarrhythmia Recorded by the Pacemakers (Intent to Treat Cohort)
Time Frame: At 2-year follow-up
Population: Intent to Treat Cohort with data available
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 90 | 96
minutes per day | 56.47 (22.61) | 24.11 (14.99)
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.2257, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Incidence of Atrial Tachyarrhythmia Recorded by the Pacemakers (Per Protocol Cohort)
Time Frame: At 2-year follow-up
Population: Per Protocol Cohort with data available
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 98 | 60
minutes per day | 40.98 (20.04) | 6.66 (4.29)
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.5480, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Incidence of Atrial Tachyarrhythmia Recorded by the Pacemakers (Intent to Treat Cohort)
Time Frame: At 5-years follow-up (study extension)
Population: Intent to Treat Cohort with data available
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 50 | 58
minutes per day | 17.73 (11.95) | 63.83 (36.82)
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.8868, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Incidence of Atrial Tachyarrhythmia Recorded by the Pacemakers (Per Protocol Cohort)
Time Frame: At 5-year follow-up (study extension)
Population: Per Protocol Cohort with data available
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 59 | 32
minutes per day | 62.75 (36.21) | 18.61 (16.61)
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.6151, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Worsening of Heart Failure
Description: Worsening of heart failure can be defined as:
  1. Heart failure-related hospitalization requiring intravenous heart failure therapy, or
  2. Emergency department visit for heart failure requiring intravenous heart failure therapy, or
  3. Any other visit in which the patient presents with signs or symptoms consistent with heart failure or heart failure exacerbation or marked decline in ejection fraction <35%, and intravenous heart failure therapy is required or titrate therapy.
  4. CRT-P or CRT-D upgrade.
Time Frame: At 5-year follow-up (study extension)
Measure: Number; unit: episodes
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 78 | 81
episodes | 19 | 17

8. Secondary Outcome: All Cause Mortality
Time Frame: At 5-year follow-up (study extension)
Measure: Number; unit: participants
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 78 | 81
participants | 14 | 11

9. Secondary Outcome: Incidence of Stroke
Time Frame: At 5-year follow-up (study extension)
Measure: Number; unit: participants
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 78 | 81
participants | 5 | 6

10. Secondary Outcome: Brain Natriuretic Peptide Levels (Intent to Treat Cohort)
Time Frame: At 2-year follow-up
Population: Intent to Treat Cohort with data available
Measure: Median (Full Range); unit: picograms per milliliter
Groups:
- RV High Septum: RV lead placement site: Patients randomised to RV high septal lead placement site (Intent to trat cohort)
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 72 | 71
picograms per milliliter | 138.2 [0.3 to 1428] | 111.3 [0.3 to 1536]
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.0525, t-test, 2 sided

11. Secondary Outcome: Brain Natriuretic Peptide Levels (Per Protocol Cohort)
Time Frame: At 2-year follow-up
Population: Per Protocol Cohort with data available
Measure: Median (Full Range); unit: picograms per milliliter
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 72 | 48
picograms per milliliter | 176.6 [0.3 to 1428] | 110.8 [0.3 to 1429]
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.1852, t-test, 2 sided

12. Secondary Outcome: Echocardiographic Measures of Left Ventricular Dyssynchrony
Description: No analysis has been done for this section since that variable was not collected during the study.
Time Frame: At 2-year follow-up
Population: No analysis has been done for this section since that variable was not collected during the study
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: 6 Minute Hall-Walk Distance (Intent to Treat Cohort)
Time Frame: At 2-year follow-up
Population: Intent to Treat Cohort with data available
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 67 | 68
meters | 391 [307 to 475] | 395 [320 to 463.25]
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.9719, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: 6 Minute Hall-Walk Distance (Per Protocol Cohort)
Time Frame: At 2-year follow-up
Population: Per Protocol Cohort with data available
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | RV Apex | RV High Septum
Number analyzed (Participants) | 68 | 47
meters | 385.5 [304.5 to 477.5] | 426.5 [355.5 to 480]
Statistical Analysis 1: Comparison: RV Apex vs RV High Septum; Test type: Superiority or Other; p = 0.8779, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | RV Apex | RV High Septum
Serious Adverse Events (participants affected / at risk) | 78/120 | 81/120
Other Adverse Events (participants affected / at risk) | 6/120 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RV Apex (N=120) | RV High Septum (N=120)
anemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
SOB (Cardiac disorders) | 25 (34) | 29 (50)
diabets (Endocrine disorders) | 1 (1) | 2 (3)
rectal bleeding (Gastrointestinal disorders) | 11 (12) | 7 (7)
chest pain (General disorders) | 10 (13) | 9 (9)
bile duct (Hepatobiliary disorders) | 2 (3) | 2 (2)
infection (Infections and infestations) | 3 (3) | 1 (1)
trauma (Injury, poisoning and procedural complications) | 10 (10) | 20 (23)
angiography (Investigations) | 2 (2) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
arthritis (Musculoskeletal and connective tissue disorders) | 6 (9) | 6 (6)
carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (10) | 8 (15)
stroke (Nervous system disorders) | 4 (8) | 9 (12)
urinary tract infection (Renal and urinary disorders) | 5 (5) | 3 (3)
prostate (Reproductive system and breast disorders) | 1 (1) | 2 (2)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 8 (10)
dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
bypass (Surgical and medical procedures) | 7 (10) | 5 (5)
raynaud's disease (Vascular disorders) | 11 (12) | 8 (13)
death (General disorders) | 19 (19) | 16 (16)
product issue (Cardiac disorders) | 9 (9) | 11 (15) — Adverse events related to the pacemaker (e.g., lead dislodgment or changing in threshold values). The term 'product issue' is taken from MedDRA 19.0 classification.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RV Apex (N=120) | RV High Septum (N=120)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No